CLINICAL TRIAL: NCT01335776
Title: An Objective Comparison of Cognitive Behavioral Therapy and Mindfulness-based Stress Reduction for the Treatment of Insomnia in Cancer Survivors Using Wrist Actigraphy: A Randomized Noninferiority Trial
Brief Title: A Comparison of MBSR and CBT for the Treatment of Insomnia in Cancer
Acronym: I-CAN SLEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Tavis S. Campbell, Associate Professor of Psychology, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RT735639
Record Dates: First submitted 2011-04-12; First posted 2011-04-14 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Cancer; Insomnia
Keywords: Mindfulness-Based Stress Reduction; Cognitive Behavior Therapy; Actigraphy; Noninferiority; MBSR; CBT-I
MeSH Terms: conditions — Neoplasms; Sleep Initiation and Maintenance Disorders | interventions — Mindfulness-Based Stress Reduction; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavior Therapy (Experimental): Cognitive Behavior Therapy for insomnia consists of stimulus control therapy, sleep restriction therapy, cognitive therapy and relaxation.
  Interventions: Behavioral: Cognitive Behavior Therapy
- Mindfulness-Based Stress Reduction (Experimental): The program consists of three primary components: theoretical material related to relaxation, meditation, and the mind-body connection; experiential practice of meditation and yoga and home based practice; group process focused on problem solving and support.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — This intervention is provided over the course of eight, weekly, 90 minute sessions, plus one 6 hour silent retreat.
  Other Names: MBSR
  Arms: Mindfulness-Based Stress Reduction
Behavioral: Cognitive Behavior Therapy — This treatment is delivered to small groups over the course of 8 weekly, 90 minute sessions
  Other Names: CBT-I
  Arms: Cognitive Behavior Therapy

SUMMARY:
Sleep disturbance in cancer patients is often overlooked despite its documented high prevalence and negative impact. There are few empirically validated non-pharmacological treatments for insomnia and many patients are unwilling to rely on sleeping medications. This study will determine whether Mindfulness-Based Stress Reduction (a program that teaches meditation and yoga) produces equivalent results with the additional benefits of reduced stress and mood disturbance, to an already established treatment for insomnia, Cognitive-Behavioral Therapy. This will allow for the expansion of treatment options for insomnia beyond what is currently available and improve quality of life for millions of cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Non metastatic cancer
* 1 month post chemotherapy/radiation treatment (hormone treatment okay)
* Diagnosis of Primary or Secondary Insomnia

Exclusion Criteria:

* Presence of another sleep disorder
* Presence of another Axis I diagnosis (not in remission)
* Inability to attend at least 5 out of the 8 treatment sessions
* Randomization Refusal
* Previous participation in CBT-I or MBSR
* Shift work

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2008-09; Primary Completion 2011-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity from baseline to 3 months | Baseline, Post-Treatment, 3 month follow up

SECONDARY OUTCOMES:
Change in objective measures of sleep using Wrist Actigraphy from baseline to 3 months | Baseline, Post Treatment, 3 month follow up
Change in subjective measures of sleep using Sleep Diaries from baseline to 3 months | Baseline (one week), During treatment (7 weeks), Post Treatment (1 week), 3 month Follow up (1 week)
Change in Pittsburgh Sleep Quality Index scores from baseline to 3 months | Baseline, Post Treatment, 3 month follow up
Change in Dysfunctional Attitudes and Beliefs about Sleep Scale scores from baseline to 3 months | Baseline, Post Treatment, 3 month folllow up
Change in Calgary Symptoms of Stress Inventory scores from baseline to 3 months | Baseline, Post Treatment, 3 month folllow up
Change in Five Facet Mindfulness Questionnaire scores from baseline to 3 months | Baseline, Post Treatment, 3 month folllow up

CONTACTS AND LOCATIONS:
Overall Officials: Tavis S Campbell, PhD, Principal Investigator — University of Calgary
Locations (1):
- Tom Baker Cancer Centre-Holy Cross Site, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811
- [Derived] Garland SN, Carlson LE, Stephens AJ, Antle MC, Samuels C, Campbell TS. Mindfulness-based stress reduction compared with cognitive behavioral therapy for the treatment of insomnia comorbid with cancer: a randomized, partially blinded, noninferiority trial. J Clin Oncol. 2014 Feb 10;32(5):449-57. doi: 10.1200/JCO.2012.47.7265. Epub 2014 Jan 6. PMID 24395850
- See also: Related Info — http://www.icansleep.ca